CLINICAL TRIAL: NCT01619462
Title: A Study of Safety and Immunogenicity of 10-valent and 13-valent Pneumococcal Conjugate Vaccines to Inform Policy Regarding Pneumococcal Vaccination of Papua New Guinean Children
Brief Title: Safety and Immunogenicity of 10-valent and 13-valent Pneumococcal Conjugate Vaccines in Papua New Guinean Children
Acronym: PCV1103
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: The University of Western Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCV1103
Record Dates: First submitted 2012-05-28; First posted 2012-06-14 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2012-09

CONDITIONS: Pneumonia; Meningitis; Bacteraemia; Sepsis; Otitis Media
Keywords: pneumococcal; vaccine; papua new guinea
MeSH Terms: conditions — Pneumonia; Meningitis; Toxemia; Sepsis; Otitis Media | interventions — 13-valent pneumococcal vaccine; PHiD-CV vaccine; 10-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synflorix or PCV10 (Other): 130 children will receive Synflorix at 1-2-3 months
  Interventions: Biological: Prevenar 13 and Synflorix
- Prevenar 13 (Other): 130 children will receive Prevenar 13 at 1-2-3 months
  Interventions: Biological: Prevenar 13 and Synflorix

INTERVENTIONS:
Biological: Prevenar 13 and Synflorix — 260 children will be randomized to receive either Prevenar 13 or Synflorix at 1-2-3 months. At 9 months 65 children in the Prevenar 13 arm and 65 children in the Synflorix arm will receive booster dose of Pneumovax and at 23 months all children will receive a micro dose of Pneumovax.Blood will be collected at 1, 4, 9, 10, 23 and 24 months to determine serotype-specific antibody responses. Nasopharyngeal swabs will also be collected to measure carriage of pneumococci and non-typeable Haemophilus influenzae.
  Other Names: Synflorix(R), PCV10; Prevenar 13(R), PCV13

SUMMARY:
The study aims to evaluate the safety and immunogenicity of the 10-valent and 13-valent pneumococcal conjugate vaccines when administered in an accelerated schedule in Papua New Guinean children, who experience early dense upper respiratory tract colonisation with a broad range of pneumococcal serotypes, and to compare antibody titres following a booster dose of polysaccharide vaccine at 9 months with those children who received no booster at the same age.

DETAILED DESCRIPTION:
The primary aim of the study is to determine whether PCV10 and PCV13 are safe and immunogenic in PNG infants for the serotypes in the respective vaccines. This study is important for the following reasons:

1. There is a lack of data worldwide on immunogenicity in populations with very high early onset of dense URT carriage.
2. The EPI immunisation schedule is very accelerated in PNG (ages 1,2 and 3 months).
3. There are not data on functional antibody to PCVs in PNG.
4. There are no data on NTHi Protein D antibody responses in PNG and worldwide in population with very high URT carriage rates from a young age, i.e. those most likely to benefit from a vaccine including NTHi protein carrier.
5. It is important to investigate impact of vaccine on carriage density in view of our finding of limited impact of 7vPCV on URT carriage.
6. There is no data on antibody responses following 10v or 13v PCV to booster with PPV as young as 9 months of age (which would be the most appropriate within the current PNG EPI schedule and in the many other third world countries).
7. There is no data on antibody responses (including functional assays) to 23vPPV challenge at age 2 years after 23vPPV booster at age 9 months in children primed with PCV.
8. The broad range of serotypes causing IPD in PNG necessitates continuing consideration of 23vPPV as a potential booster at age 9 months.
9. Serotype-specific B cell memory is an important aspect that we can now test to address immunological safety of PPV in children primed with PCV.
10. The Global Alliance for Vaccines and Immunisation (GAVI) and the World Health Organisation (WHO) have committed to the introduction of PCV for infants in GAVI-eligible countries (including PNG) using novel funding mechanism. In PNG, the introduction of a PCV is planned for 2013.

ELIGIBILITY:
Inclusion Criteria:

* Health infants between 28 - 35 days old

Exclusion Criteria:

* Infants of women not intending to remain in the are for at least two years
* Birth weigh < 2000 g (2kg)
* Severe congenital abnormalities
* Mother or child known to be HIV positive

Ages: 28 Days to 35 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-04 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of children with serotype-specific IgG concentration >= 0.35ug/ml at 4 and 9 months of age for 90% of PCV vaccine serotypes and proportion of children with OPA >=1:8 titres at 4, 10 and 24 months | 3 years
  IgG concentration to vaccine serotypes are >= 0.35ug/ml post-dose 3 at 4 and 9 months. Serotype-specific IgG concentration >=0.35ug/ml is protective level against invasive pneumococcal diseases. Opsonophagocytic titre of >=1:8 examined at 4, 10 and 24 months will inform on functional antibodies induced by vaccination.

SECONDARY OUTCOMES:
Compare antibody concentrations to pneumococcal and Haemophilus influenzae protein antigens. | 2 years
  Measure antibody titres to surface proteins of pneumococci and Hi including Hi protein D, the carrier protein in PCV10 (Synflorix).
Determine carriage rates and bacterial load of pneumococci and H.influenzae | 3 years
  Proportion of carriage before and after vaccination will be measured using conventional culture methods. Bacterial load will be measured using PCR to determine impact of vaccines
Determine rates of hospital admission for acute respiratory tract infections at 9 and 23 months | 2 yrs
  Admissions and morbidity for acute respiratory tract infections will be documented at 9 and 23 months.

CONTACTS AND LOCATIONS:
Overall Officials: William S Pomat, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research; Deborah Lehmann, MSc, Principal Investigator — Telethon Institute for Child Health Research; Peter Richmond, MD, Principal Investigator — The University of Western Australia
Locations (1):
- Papua New Guinea Institute of Medical Research, Goroka, Eastern Highlands Province, Papua New Guinea

REFERENCES:
- [Derived] Orami T, Aho C, Ford RL, Pomat WS, Greenhill A, Kirkham LA, Masiria G, Nivio B, Britton KJ, Jacoby P, Richmond PC, van den Biggelaar AHJ, Lehmann D. Pneumococcal carriage, serotype distribution, and antimicrobial susceptibility in Papua New Guinean children vaccinated with PCV10 or PCV13 in a head-to-head trial. Vaccine. 2023 Aug 23;41(37):5392-5399. doi: 10.1016/j.vaccine.2023.07.026. Epub 2023 Jul 20. PMID 37479616
- [Derived] Martinovich KM, Rahman T, de Gier C, Seppanen EJ, Orami T, Granland CM, Francis J, Yoannes M, Corscadden KJ, Ford R, Jacoby P, van den Biggelaar AHJ, Bakaletz LO, Cripps AW, Lehmann D, Richmond PC, Pomat WS, Kirkham LS, Thornton RB. Differences in Pneumococcal and Haemophilus influenzae Natural Antibody Development in Papua New Guinean Children in the First Year of Life. Front Immunol. 2021 Aug 10;12:725244. doi: 10.3389/fimmu.2021.725244. eCollection 2021. PMID 34447389
- [Derived] Rahman T, de Gier C, Orami T, Seppanen EJ, Granland CM, Francis JP, Michael A, Yoannes M, Corscadden KJ, Ford RL, Martinovich KM, Jacoby P, van den Biggelaar AHJ, Lehmann D, Richmond PC, Pomat WS, Thornton RB, Kirkham LS. PCV10 elicits Protein D IgG responses in Papua New Guinean children but has no impact on NTHi carriage in the first two years of life. Vaccine. 2021 Jun 11;39(26):3486-3492. doi: 10.1016/j.vaccine.2021.05.022. Epub 2021 May 21. PMID 34024658
- [Derived] Pomat WS, van den Biggelaar AHJ, Wana S, Francis JP, Solomon V, Greenhill AR, Ford R, Orami T, Passey M, Jacoby P, Kirkham LA, Lehmann D, Richmond PC; 10v13v PCV Trial Team. Safety and Immunogenicity of Pneumococcal Conjugate Vaccines in a High-risk Population: A Randomized Controlled Trial of 10-Valent and 13-Valent Pneumococcal Conjugate Vaccine in Papua New Guinean Infants. Clin Infect Dis. 2019 Apr 24;68(9):1472-1481. doi: 10.1093/cid/ciy743. PMID 30184183
- [Derived] Lehmann D, Kirarock W, van den Biggelaar AHJ, Passey M, Jacoby P, Saleu G, Masiria G, Nivio B, Greenhill A, Orami T, Francis J, Ford R, Kirkham LA, Solomon V, Richmond PC, Pomat WS; 10v13v PCV trial team. Rationale and methods of a randomized controlled trial of immunogenicity, safety and impact on carriage of pneumococcal conjugate and polysaccharide vaccines in infants in Papua New Guinea. Pneumonia (Nathan). 2017 Dec 25;9:20. doi: 10.1186/s41479-017-0044-z. eCollection 2017. PMID 29299402